CLINICAL TRIAL: NCT05014607
Title: Personalized Multi-peptide Vaccination in Combination With the TLR1/2 Ligand XS15 in Cancer Patients
Acronym: InHeVac01
Status: Available | Type: Expanded Access
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: InHeVac01
Record Dates: First submitted 2021-07-23; First posted 2021-08-20 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Expanded Access Types: Individual, Intermediate

INTERVENTIONS:
Biological: Personalized multi-peptide vaccine — Peptide vaccine: Personalized multi-peptide vaccine cocktails consisting of 200-300µg each of 1-10 tumor-associated peptides selected individually based on the patient-individual HLA allotypes and HLA ligandome analysis of tumor cells Peptides are synthesized in the GMP-certified Wirkstoffpeptidlabor at the University of Tübingen and will be formulated at the GMP-Center of the University Hospital Tübingen.
  Peptides will be administered subcutaneously (s.c.) together with the TLR1/2 ligand XS15 emulsified in Montanide ISA 51 VG as adjuvant.
  Vaccination will take place every 6 weeks. A total of two to five vaccinations are planned.
  Treatment schedule:
  Vaccination will take place every 6 weeks. A total of two to five vaccinations are planned, depended on the induction of peptide-specific T-cell responses.
  Other Names: Adjuvants XS15 and Montanide ISA 51 VG

SUMMARY:
The aim of this project is to provide personalized multi-peptide vaccination in combination with the TLR1/2 ligand XS15 to individual patients with advanced solid and hematological malignancies without any approved treatment options.

DETAILED DESCRIPTION:
Ethics: Patient treatment will be conducted according to §13 Absatz 2b, AMG.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of advanced malignant disease
* Advanced malignant disease without any available standard of care treatment option
* Low tumor cell burden
* Live expectancy > 6 month
* Ability to understand and voluntarily sign an informed consent form.
* Ability to adhere to the study visit schedule and other protocol requirements
* Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 2.

Exclusion Criteria:

* Pregnant or lactating females.
* Treatment regimens inducing sever T cell deficiencies
* Treatment-related side effect > CTC grade 2 (CTCAE V5.0
* Participation in any clinical study or having taken any investigational therapy, which would interfere with the studys primary and secondary end points within 2 weeks prior to vaccination
* Pre-existing auto-immune disease except for Hashimoto thyroiditis and mild (not requiring immunosuppressive treatment) psoriasis

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Helmut R Salih, MD, Study Chair — CCU Translational Immunology, University Hospital Tübingen, Germany

REFERENCES:
- See also: Department CCU Translational Immunology — https://www.medizin.uni-tuebingen.de/en-de/das-klinikum/einrichtungen/kliniken/medizinische-klinik/kke-translationale-immunologie